CLINICAL TRIAL: NCT02267746
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Vehicle-Controlled Study to Evaluate the Safety and Therapeutic Equivalence of a Generic Tazarotene Foam 0.1%(Actavis) and the Reference Listed Fabior™(Tazarotene Foam, 0.1%) (Stiefel Laboratories, Inc.) in Treatment of Subjects With Acne Vulgaris
Brief Title: A Study To Evaluate The Safety And Therapeutic Equivalence of Tazarotene Foam 0.1% in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WAT 14-1096
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Results first posted 2020-05-11 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fabior™(tazarotene) (Active Comparator): Reference listed drug: Fabior™ 0.1% foam (Stiefel)
  Interventions: Drug: Tazarotene (Fabior™)
- Tazarotene (Experimental): Tazarotene 0/1% foam (Actavis)
  Interventions: Drug: Tazarotene (Actavis)
- Vehicle foam (Placebo Comparator): Foam vehicle of the test product (Actavis)
  Interventions: Drug: Vehicle foam

INTERVENTIONS:
Drug: Tazarotene (Fabior™)
  Arms: Fabior™(tazarotene)
Drug: Tazarotene (Actavis)
  Arms: Tazarotene
Drug: Vehicle foam
  Arms: Vehicle foam

SUMMARY:
The purpose of this study is to compare the safety and therapeutic equivalence of a generic tazarotene foam 0.1% and the reference listed Fabior™ (tazarotene foam, 0.1%) in the treatment of acne vulgaris.

DETAILED DESCRIPTION:
Although topical retinoids have been individually used to successfully treat acne vulgaris, Fabior™ (Tazarotene) Foam, 0.1% is a safe and effective topical therapy used for the treatment of acne vulgaris. Actavis has developed a generic formulation of Tazarotene Foam, 0.1%, and the current study is designed to evaluate the safety and efficacy of this formulation.

ELIGIBILITY:
Inclusion Criteria:

Healthy male or nonpregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris.

Informed Consent/Assent: Subjects ages 12 to 17 years inclusive must have provided IRB approved written assent; this written assent must be accompanied by an IRB approved written informed consent from the Subject's legally acceptable representative (i.e., parent or guardian). In addition, all Subjects or their legally acceptable representatives (i.e., parent or guardian) must sign a HIPAA authorization.

Subjects must have a minimum ≥ 30 non-inflammatory lesions (i.e., open and closed comedones) AND ≥ 25 inflammatory lesions (i.e., papules and pustules) AND no cystic lesions and only up to 1 facial nodular lesion (less than or equal to 5 mm) on the face. For the purposes of study treatment and evaluation, these lesions should be limited to the facial treatment area excluding the eyes, the lips, and angles of the nose (i.e. the lines around the nostrils and under the nostrils) and all mucus membranes. Subjects may have acne lesions on other areas of the body which will also be excluded from the count, treatment, and the Investigator's Global Assessment (IGA) evaluation (e.g., on the back, chest and arms).

Subjects must have a severity grade 3, or 4 as per the Investigator's Global Assessment (IGA) (Section 6.2).

Subjects must be willing to refrain from using all other topical acne medications or antibiotics during the 12-week treatment period for acne vulgaris, other than the Investigational Product.

Female Subjects of childbearing potential (excluding women who are surgically sterilized or postmenopausal for at least 1 year), must have a negative urine pregnancy test (with sensitivity down to at least 50mIU/ml hCG) within 2 weeks prior to baseline.

Female Subjects of childbearing potential (excluding women who are surgically sterilized or postmenopausal for at least 1 year), must be willing to use an acceptable form of birth control from the day of the first dose administration.. For the purpose of this study the following are considered acceptable methods of birth control: oral or injectable contraceptives, contraceptive patches, Depo-Provera® (stabilized for at least 3 months); NuvaRing® (vaginal contraceptive); Implanon™ (contraceptive implant) double barrier methods (e.g. condom and spermicide); IUD, or abstinence with a 2nd acceptable method of birth control should the Subject become sexually active. A sterile sexual partner is NOT considered an adequate form of birth control.

All male Subjects must agree to use accepted methods of birth control with their partners, from the day of the first dose administration. Abstinence is an acceptable method of birth control for males.

Subjects must be willing and able to understand and comply with the requirements of the protocol, including attendance at the required study visits.

Subjects who use make-up must have used the same brands/types of make-up for a minimum period of 14 days prior to study entry and must agree to not change make-up brand/type or frequency of use throughout the study.

-

Exclusion Criteria:

Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.

Subjects with a history of hypersensitivity or allergy to tazarotene and its excipients, and/or any of the study medication ingredients.

Subjects with the presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris. Such conditions include, but are not limited to the following: auto immune disease, rosacea; seborrheic dermatitis; perioral dermatitis; corticosteroid-induced acne; carcinoid syndrome; mastocytosis; acneform eruptions caused by make-up, medication, facial psoriasis and facial eczema, squamous cell carcinoma, steroid folliculitis, or bacterial folliculitis).

Subjects who have acne congoblata, acne fulminans, and secondary acne (e.g., chloracne and drug induced acne) will be excluded from participation.

Subjects with excessive facial hair (e.g. beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of acne vulgaris.

Subjects who have used any of the following within 6 months prior to baseline or use during the study:

1. oral retinoids (e.g. Accutane®)
2. therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).

Subjects who have used estrogens or oral contraceptives for less than 3 months prior to baseline; use of such therapy must remain constant throughout the study.

Subjects who use androgen receptor blockers (such as spironolactone or flutamide) will be excluded from study participation.

Subjects who have had cosmetic procedures (e.g., facials, wax depilation) which may affect the efficacy and safety profile of the investigational product within 14 days prior to study entry. Cosmetic procedures and facials are prohibited throughout the study.

Subjects who have received radiation therapy and/or anti-neoplastic agents within 90 days prior to baseline.

Subjects who have had laser therapy, electrodessication and phototherapy (e.g., ClearLight®) to the facial area within 180 days prior to study entry.

Subjects who have used any of the following procedures on the face within 1 month prior to baseline or during the study:

1. cryodestruction or chemodestruction,
2. dermabrasion,
3. photodynamic therapy,
4. acne surgery,
5. intralesional steroids, or
6. X-ray therapy.

Subjects who have used any of the following treatments within 1 month prior to baseline or during the study:

1. systemic corticosteroids (including intranasal and inhaled corticosteroids)
2. systemic antibiotics,
3. systemic treatment for acne vulgaris (other than oral retinoids which need a 6-month washout), or
4. systemic anti-inflammatory agents.

Subjects who have used any of the following treatments within 14 days prior to baseline or during the study:

1. topical steroids,
2. topical retinoids including over-the-counter preparations,
3. α-hydroxy/glycolic acid
4. topical anti-inflammatory agents, or
5. topical antibiotics.

Subjects who have started hormonal therapy or changed the dosage of their hormonal therapy within 3 months prior to baseline will be excluded from study participation. The dosage and frequency of use of any hormonal therapy started greater than 3 months prior to baseline must remain unchanged throughout the study (Visit 1 through Visit 4). Hormonal treatments include, but are not limited to, estrogenic and progestational agents such as birth control pills.

Subjects who have unstable medical disorders that are clinically significant or life-threatening diseases will be excluded from study participation.

Subjects with current facial sunburn at baseline or subjects who will have excessive use of tanning booths, sunbathing, or excessive exposure to the sun during the study.

Subjects who will engage in activities that involve excessive or prolonged exposure to sunlight or weather extremes, such as wind or cold.

Subjects who have on-going malignancies requiring systemic treatment will be excluded from study participation. In addition, Subjects who have any malignancy of the skin of the facial area will be excluded.

Subjects who consume excessive amounts of alcohol (greater than two drinks per day) or use drugs of abuse (including, but not limited to cannabinoids, cocaine and barbiturates).

Subjects who have had general anesthesia for any reason and subjects who have received neuromuscular blocking agents within 14 days prior to study entry will be excluded from study participation.

Subjects who have participated in an investigational drug study (i.e., Subjects have been treated with an Investigational Drug) within 30 days prior to baseline will be excluded from study participation. Subjects who are participating in non-treatment studies such as observational studies or registry studies can be considered for inclusion.

Subjects who have been previously enrolled in this study.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 893 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keri Winkler, Study Director — Akesis, LLC
Locations (14):
- United States (13):
  - Encino, California
  - Center for Dermatology Clinical Research, Fremont, California
  - Moore Clinical Research, Brandon, Florida
  - LCC Medical Research Institute, Miami, Florida
  - International Dermatology Research, Miami, Florida
  - FXM Research Corp, Miami, Florida
  - FXM Research Miramar, Miramar, Florida
  - Moore Clinical Research, Tampa, Florida
  - Atlantic Clinical Research Collaborative, Wellington, Florida
  - Omega Medical Research, Warwick, Rhode Island
  - Research Across America, Dallas, Texas
  - Research Across America, Plano, Texas
  - Dermatology Research Center, Salt Lake City, Utah
- FXM International, Belize City, Belize

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 893 subjects were randomized and analyzed; 869 qualified for the mITT population and 758 for the PP population.
Groups:
- Test: Tazarotene 0.1% foam (Actavis LLC)
- Reference: Reference listed drug: Fabior™ 0.1% (tazarotene) foam (Stiefel Laboratories LLC)
- Vehicle: Vehicle foam of the test product (Actavis LLC)
Period: Overall Study
Arm/Group | Test | Reference | Vehicle
Started | 298 | 296 | 299
Completed | 277 | 274 | 278
Not Completed | 21 | 22 | 21
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Protocol Violation | 8 | 7 | 3
Not completed — Lack of Efficacy | 11 | 11 | 15
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Miscellaneous | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 874 (97.9%) of the 893 randomized subjects applied study treatment during the baseline visit, and were therefore retained in the Safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Reference | Vehicle | Total
Number analyzed (Participants) | 292 | 288 | 294 | 874
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.5 (7.76) | 21.1 (7.26) | 21.0 (7.03) | 21.2 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 107 | 107 | 327
  Male | 179 | 181 | 187 | 547
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 118 | 110 | 115 | 343
  Not Hispanic or Latino | 174 | 178 | 179 | 531
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 6 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 3
  Black or African American | 109 | 116 | 91 | 316
  White | 177 | 160 | 193 | 530
  More than one race | 1 | 5 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Inflammatory (Papules and Pustules) Lesion Counts
Description: For the purposes of study treatment and evaluation, these lesions were limited to the facial treatment area excluding the eyes, the lips, and angles of the nose (i.e., the lines around the nostrils and under the nostrils) and all mucus membranes.
Time Frame: Mean percent change from baseline to Week 12
Population: Mean percent change from baseline to Week 12 in Per Protocol Population
Measure: Mean (Standard Deviation); unit: Percent change in inflammatory lesions
Groups:
- Vehicle: Placebo foam (Actavis LLC)
Arm/Group | Test | Reference | Vehicle
Number analyzed (Participants) | 187 | 185 | 195
Percent change in inflammatory lesions | -48.25 (26.743) | -52.72 (22.792) | -45.03 (24.092)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — Estimates of mean percent change from baseline were calculated (separately for inflammatory and non-inflammatory lesions) for the Test and Reference treatment, and then the 90% confidence interval (CI) for the mean ratio was constructed using Fieller's method; Mean Difference (Net) = 0.93, 90% CI 2-sided [0.86 to 1.02] — Therapeutic equivalence was established if the 90% CIs for the ratio of Test/Reference means, for both lesion types, were contained within the interval [0.80, 1.25] for the PP population

2. Primary Outcome: Percent Change in the Non-inflammatory (Open and Closed Comedones) Lesion Counts
Description: Estimates of mean percent change from baseline for non-inflammatory lesions for the Test and Reference treatment.
Time Frame: Mean percent change from baseline to Week 12
Population: Percent change in the non-inflammatory lesions in Per Protocol Population.
Measure: Mean (Standard Deviation); unit: percent change in noninflammatory lesion
Groups:
- Vehicle Foam: Placebo Foam (Actavis LLC)
Arm/Group | Test | Reference | Vehicle Foam
Number analyzed (Participants) | 187 | 185 | 195
percent change in noninflammatory lesion | -41.98 (21.125) | -44.51 (20.062) | -37.42 (24.126)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.96, 90% CI 2-sided [0.89 to 1.04] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: The Proportion of Subjects With an IGA Score That is at Least 2 Grades Less Than the Baseline Assessment
Time Frame: IGA score at Week 12 compared to baseline
Population: Treatment success based on IGA score at Week 12 in PP population
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference | Vehicle
Number analyzed (Participants) | 252 | 247 | 259
Participants
  Success | 103 | 119 | 88
  Failure | 149 | 128 | 171
Statistical Analysis 1: Comparison: Test vs Reference; Success was defined as an IGA score at Week 12 that was at least two grades less than the baseline assessment. Failure was defined as an IGA score that was the same, higher, or one grade lower than the baseline assessment; Test type: Equivalence — Therapeutic equivalence was established if the 90% CI for the difference was contained within the interval [-0.20, +0.20] for PP population; Mean Difference (Net) = -0.073, 90% CI 2-sided [-0.150 to 0.004] — Therapeutic equivalence was established if the 90% CI for the difference was contained within the interval [-0.20, +0.20] for the PP population

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over approximately 13 weeks.
Arm/Group | Test | Reference | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/292 | 0/288 | 0/294
Serious Adverse Events (participants affected / at risk) | 0/292 | 0/288 | 0/294
Other Adverse Events (participants affected / at risk) | 41/292 | 55/288 | 43/294
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=292) | Reference (N=288) | Vehicle (N=294)
Eye Pain (Eye disorders) | 0 | 0 | 1
Eye Pruritis (Eye disorders) | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 0
Oral pain (Gastrointestinal disorders) | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Application site reaction (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Cyst (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 1
Food allergy (Immune system disorders) | 0 | 1 | 0
Influenza (Infections and infestations) | 4 | 5 | 5
Localized infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 7 | 5 | 9
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 12 | 17 | 20
Migraine (Nervous system disorders) | 0 | 1 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 7 | 3 | 5
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed